CLINICAL TRIAL: NCT05202977
Title: A Prospective，Multicenter, Single-arm Clinical Trial to Evaluate Safety and Efficacy of SinocrownTM Transcatheter Aortic Valve Replacement System With Accessories in Patients With Symptomatic, Calcified and Severe Aortic Stenosis
Brief Title: Safety and Efficacy of SinocrownTM Transcatheter Aortic Valve Replacement System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-TAVR-2021
Record Dates: First submitted 2021-12-31; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SinocrownTM Transcatheter Aortic Valve Replacement System (Experimental): The experimental apparatus consisted of artificial aortic valve, transporter and grip-loading system.
  Interventions: Device: SinocrownTM Transcatheter Aortic Valve Replacement System

INTERVENTIONS:
Device: SinocrownTM Transcatheter Aortic Valve Replacement System — Subjects receiving SinocrownTM Transcatheter Aortic Valve Replacement System of Lepu Medical

SUMMARY:
This study was designed to preliminary verify the safety and of efficacy of SinocrownTM Transcatheter Aortic Valve Replacement System With accessories in patients with symptomatic, calcified and severe aortic stenosis using objective performance criteria

DETAILED DESCRIPTION:
This prospective, single-center, single-arm clinical trial was designed to preliminary confirm the safety and efficacy of SinocrownTM transcatheter aortic valve system with accessories.

According to the inclusion and exclusion criteria, 10 patients were enrolled and implanted with SinocrownTM .Patients will been followed up 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years after valve implantation. The main follow-up included clinical symptoms and signs, cardiac ultrasound, etc. The primary endpoint was device success after TAVR, Secondary endpoints included procedural success, all-cause mortality, myocardial infarction, disabling stroke, severe bleeding, acute kidney injury, permanent pacemaker implantation, vascular complications, other complication, MACCEs, valvular function , cardiac function improvement, quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years ;
2. Autologous degenerative aortic stenosis（evaluated by echocardiography: transaortic valve pressure gradient ≥40mmHg , or transaortic valve blood flow rate ≥4m/s, or aortic Valve area<1.0cm2, or AVA <0.5cm2 /m2）
3. Patients with aortic annulus size≥17.5mm and ≤29mm (echocardiography measurement);
4. The diameter of the ascending aorta of the patient was < 45mm.
5. Appear obvious symptoms caused by aortic stenosis, NYHA class Ⅱ to IV;
6. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
7. Subjects are willing to accept all clinical follow-up.
8. The cardiologist and cardiac surgeon evaluated the subject as unsuitable for surgical treatment (the risk of death or irreversible complications within 30 days after operation is expected to be above 50% , or contraindicated comorbidities such as prior chest radiotherapy, liver failure, diffuse severe calcification of the aorta, extreme weakness, etc.). Or Moderate or higher surgical risk (STS score ≥ 4%).

Exclusion Criteria:

1. defined as Q-wave myocardial infarction or non-Q-wave myocardial infarction with CK-MB level ≥ 2 times the upper limit of normal value and / or Tn increase.
2. Subjects with congenital unicuspid, without calcification.
3. Any therapeutic or traumatic cardiac surgery within 30 days (within 3 months in case of drug-eluting stents implantation)
4. The patient's heart has been implanted with other artificial heart valves, artificial rings, or severe mitral annulus calcification (MAC), severe (> 3 +) mitral insufficiency.
5. Hematological abnormalities, including leukopenia (WBC<3×109/L), acute anemia (HB <90g/L), thrombocytopenia (PLT<50×109/L), bleeding constitution and coagulopathy ；
6. Subjects with hemodynamic instability, requiring continuous mechanical heart assistance.
7. Subjects who need emergency surgery for any reason;
8. Hypertrophic cardiomyopathy with or without obstruction;
9. Severe left ventricular dysfunction, left ventricular ejection fraction (LVEF) <20%;
10. The echocardiogram indicates the presence of a thrombus or vegetation;
11. A history of active peptic ulcer or upper gastrointestinal bleeding within 3 months;
12. Are allergic to nickel titanium alloys or contrast agents, and cannot tolerate anticoagulation and antiplatelet therapy;
13. Cerebrovascular accident occurred within 6 months, including transient ischemic attack;
14. renal insufficiency(creatinine> 3.0mg/dL) and/or end-stage renal disease requiring Renal dialysis;
15. Life expectancy< 12 months;
16. Significant aortic diseases, including abdominal aortic or thoracic aortic aneurysm(defined as maximum lumen diameter > 50mm, obvious distortion), atherosclerosis of the aortic arch(especially bulge with thickness > 5mm or ulceration), narrowing of the abdominal or thoracic aorta(especially calcification and irregular surface), and severe curvature of the thoracic aorta;
17. The iliac-femoral artery cannot be inserted with a guide sheath of 22F or above, such as severely obstructed with calcification, severely tortuous or vessel diameter less than 6mm;
18. Screening participant who is participating in other drug or medical device clinical trials;
19. Active infective endocarditis or other active infections;
20. Anatomically, the approach or aortic root is not suitable for TAVR (such as a high risk of coronary artery occlusion).
21. Other conditions considered by the investigator to be inappropriate for participation in this clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
device success | immediate post-surgical
  Immediate postoperative device success was defined as : successfully loading the valve into the delivery system, sending it to the target site through the delivery system, accurately releasing the artificial aortic valve and completely withdrawing the delivery system (valve orifice area > 1.2cm2, mean aortic gradient< 20mmhg or maximal aortic valve velocity < 3 m/ s, and there is no moderate or severe valve stenosis)

SECONDARY OUTCOMES:
Procedural success | immediate post-surgical
  Device success without death and aortic valve reintervention during operation
All-cause mortality | immediate post-surgical, 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  including cardiac, non-cardiac and unexplained deaths
Myocardial infarction | immediate post-surgical, 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Rate of patients with myocardial infarction
Rate of disabling stroke | 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Disabling stroke was defined as mRS ≥ 2, and the mRS score increased by more than 1 point compared with the last visit
Rate of Severe bleeding(life-threatening or disabling) | 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Severe degree was defined as type 3a or above（according to BARC）
acute kidney injury | 7 days after procedure/prior to discharge, 30 days after procedure
  Rate of patients with acute kidney injury
permanent pacemaker implantation | 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Rate of patients implanted with permanent pacemaker
vascular complications | immediate post-surgical, 7 days after procedure/prior to discharge
  Vascular complications mainly include dissection, occlusion, rupture and bleeding of access vessels.
other operative complication | immediate post-surgical, 7 days after procedure/prior to discharge
  including conversion to surgery, unexpected cardiopulmonary mechanical assistance, coronary artery occlusion, ventricular septal perforation, mitral valve injury or loss of function, pericardial tamponade, endocarditis, valve thrombosis, valve ectopic (displacement, embolization, misrelease), and so on.
The incidence of major adverse cardiovascular and cerebrovascular events during the trial(MACCEs) | immediate post-surgical, 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years
  Incidence of MACCEs (including mortality, stroke, myocardial infarction, reoperation, arrhythmias and conduction blocks) during the trial.
Valve and heart function | immediate post-surgical, 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months
  Doppler echocardiography was used to evaluate the valve performance at each follow-up point, including valve orifice area, mean aortic gradient, degree of valve regurgitation, left ventricular ejection fraction LVEF, end diastolic left ventricular inner diameter LVEDd, moderate or above perivalvular leakage PVL, and degree of aortic stenosis.
Cardiac function improvement | 7 days after procedure/prior to discharge, 30 days, 6 months, 12 months
  Cardiac function improvement is accessed by NYHA cardiac function classification increases from baseline to discharge, 30 days, 6 months, 12 months
Quality of life of patients | 30 days, 6 months, 12 months
  Quality of Life of patients accessed by EuroQol-5 Dimensions (EQ-5D) Questionnaire. The higher scores mean a better health state. Recording changes from baseline to 30 days, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Wu, Study Chair — Heifei High-tech Cardiovascular hospital; Weiyi Fang, Study Chair — Heifei High-tech Cardiovascular hospital
Locations (1):
- Hefei High-tech Cardiovascular hospital, Hefei, Anhui, China